CLINICAL TRIAL: NCT00907400
Title: Phase I, Open-label, Randomized, 2-way Crossover Study to Assess Relative Bioavailability of Single Oral Dose of Naproxen as PN400 Compared to Naproxen as Naprosyn E Under Fasting and Fed Conditions in Healthy Volunteers
Brief Title: Phase I Study to Evaluate Bioavailability of Naproxen as PN400 Compared to Naproxen as Naprosyn E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Sostek, MD, Medical Science Director, Development Projects, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D1120C00024; EudraCT No 2009-011738-87
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Phase 1; Healthy Volunteer; Healthy Volunteer Study
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PN400
  Interventions: Drug: PN400
- 2 (Active Comparator): Naprosyn E
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: PN400 — oral tablet
  Other Names: VIMOVO™
  Arms: 1
Drug: Naproxen — oral tablet
  Other Names: Naprosyn E
  Arms: 2

SUMMARY:
The purpose of the study is to investigate the uptake in the body of naproxen; one of the two active substances in PN400. We also want to show that the body's uptake of naproxen given as PN400 is comparable to that of currently marketed naproxen tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18-55 yrs. of age (inclusive) at Screening Visit
* Body Mass Index (BMI) of greater than or equal to 19 to less than or equal to 30 kg/m2 and weight of greater than or equal to 50 to less than or equal to 100 kg
* Clinically normal physical exams and laboratory measurements

Exclusion Criteria:

* Subject has received another investigational drug within 4 weeks preceding this study or planning to participate in another study at any time during the period of this study
* Any significant medical or psychiatric condition that could affect the interpretation of the PK data, or which otherwise would contraindicate participation in a clinical trial
* Any GI disease, abnormality or gastric surgery that may interfere with gastric emptying, motility and drug absorption
* Subject who has donated a unit of blood or plasma within 3 months prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | pre-dose and multiple times post-dose

SECONDARY OUTCOMES:
Safety | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, MD, Study Director — AstraZeneca; Aslak, Rautio, MD, Principal Investigator — Quintiles Hermelinen; Elisabeth Eden, MD, Principal Investigator — Quintiles AB
Locations (2):
- Sweden (2):
  - Research Site, Luleå
  - Research Site, Uppsala